CLINICAL TRIAL: NCT04249427
Title: A Randomized, Double-Blinded, Single Site Study to Evaluate the Efficacy of Erenumab for Treatment of Idiosyncratic Facial Pain Mimicking Rhinosinusitis
Brief Title: Erenumab for Idiosyncratic Facial Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: David Jang, M.D. (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, David Jang, M.D., Associate Professor of Head and Neck Surgery and Communication Sciences, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00104284
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Facial Pain; Rhinosinusitis
MeSH Terms: conditions — Facial Pain; Rhinosinusitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erenumab (Active Comparator): 140mg Erenumab administered by subcutaneous injection (in the abdomen, thigh, or upper arm), once monthly for six months.
  Interventions: Drug: Erenumab Prefilled Syringe
- Placebo (Placebo Comparator): Placebo administered by subcutaneous injection (in the abdomen, thigh, or upper arm), once monthly for six months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Erenumab Prefilled Syringe — 140mg Erenumab, pre-filled syringe given by subcutaneous injection
  Arms: Erenumab
Other: Placebo — Placebo, pre-filled syringe given by subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a phase IV randomized, double-blinded, placebo-controlled study to evaluate the efficacy of Erenumab in subjects with midfacial pain or pressure, without clinical or radiographic evidence of sinusitis.

DETAILED DESCRIPTION:
Eligible participants are randomized to receive either Erenumab or placebo by subcutaneous injection once monthly for 6 months. Study duration is eight months which includes a 30 day screening/lead-in period and 6 monthly treatment visits followed by a follow-up visit one month following the last dose of study drug administration. Participants will be expected to score on a scale of 1 to 10 their symptoms of facial pain/pressure, nasal congestion, and rhinorrhea as well well as any rescue medicines taken for pain each day via a mobile app.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age and older presenting to Duke Head & Neck Surgery and Communications Sciences clinic for evaluation of rhinosinusitis and/or facial pain or pressure.
2. Symptoms are present at least 10 days a month for the last 3 months as reported by subject.
3. Symptoms must include midfacial pain or uncomfortable pressure (may be unilateral or bilateral), which is defined as pain in the regions overlying the maxillary, ethmoid, frontal sinuses either together or individually.
4. Nasal endoscopy in the last three months shows no signs of inflammation (i.e. thick drainage, polyps, watery edema in the middle meatus or spheno-ethmoid recess (mild edema permitted).
5. Sinus CT scan or MRI within 12 months of enrollment during a symptomatic period shows no more than scattered minimal mucosal edema or mucous retention cyst with patent infundibula bilaterally. For subjects with a CT scan more than 12 months old or just an MRI, a CT will be repeated for study purposes. For patients with CT scans less than 12 months old, a CT will be repeated for study purposes if the subject has changes in symptoms suggestive of sinusitis.
6. Ability to read/write English.
7. Has a smart phone, ipod or iPad touch for completion of the EMA on a daily basis.

Exclusion Criteria:

1. Hypersensitivity to erenumab or to any of the drug components (acetate, polysorbate, and sucrose).
2. Previous exposure to erenumab or any other CGRP inhibitor in the six months prior to treatment.
3. Allergy to latex.
4. Inability to differentiate facial pain from other headaches.
5. Non-English speaking or unable to provide written informed consent.
6. On a preventative migraine medication (see below) during the 30 day lead-in period:

   * Category 1: Divalproex sodium, sodium valproate
   * Category 2: Topiramate
   * Category 3: Beta blockers (for example: atenolol, bisoprolol, metoprolol, nadolol, ebivolol, pindolol, propranolol, timolol)
   * Category 4: Tricyclic antidepressants (for example: amitriptyline, nortriptyline, protriptyline)
   * Category 5: Serotonin-norepinephrine reuptake inhibitors (for example: venlafaxine, desvenlafaxine, duloxetine, milnacipran)
   * Category 6: Flunarizine, verapamil
   * Category 7: Lisinopril, candesartan
7. Received botulinum toxin (Botox) to the head and neck for migraines in the last four months.
8. More than one major open surgery of the nose or sinuses for sinonasal cancer.
9. History of uncontrolled or unstable blood pressure.
10. History of liver failure.
11. History of metastatic malignancy in the last five years or actively undergoing treatment for cancer.
12. Active seizure disorder or other significant neurological conditions other than migraine.
13. Myocardial infarction (MI), stroke, transient ischemic attack (TIA), unstable angina, or coronary artery bypass surgery or other revascularization procedure within 12 months prior to screening.
14. History or evidence of any other unstable or clinically significant medical condition that in the opinion of the sponsor-investigator/ Principal Investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
15. Evidence of drug or alcohol abuse or dependence within 12 months prior to screening, based on medical records or patient self-report.
16. Pregnant or breastfeeding, or expecting to conceive during the study, including through 16 weeks after the last dose of investigational product or placebo
17. Female subject of childbearing potential who is unwilling to use an acceptable method of effective contraception during treatment with investigational product or placebo through 16 weeks after the last dose of investigational product. Female subjects not of childbearing potential are defined as any female who is post-menopausal by history, defined as:

    * Age ≥ 55 years with cessation of menses for 12 or more months, OR
    * Age < 55 years but no spontaneous menses for at least 2 years, OR
    * Underwent bilateral oophorectomy, bilateral salpingectomy, or hysterectomy
18. Unlikely to be able to complete all protocol required study visits or procedures.
19. Currently receiving treatment in another investigational device or drug study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jang, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center and affiliated practices, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four participants withdrew prior to administration of injection.
Period: Overall Study
Arm/Group | Erenumab | Placebo
Started | 13 | 12
Completed | 9 | 8
Not Completed | 4 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erenumab | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (11.5) | 43.2 (12.5) | 47.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Number of Days Per Month With Significant Mid-facial Pain or Pressure
Description: Significant mid-facial pain or pressure defined as greater than 4/10 on scale of 1 to 10, measured by daily diary completion. Reported as the change from baseline to six months.
Time Frame: Baseline, 1,3, and 6 months
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 13 | 12
days per month | -6.0 (6.9) | -5.8 (8.0)
Statistical Analysis 1: Comparison: Erenumab vs Placebo; Test type: Equivalence — Test if the change in mean number of days with significant mid-facial pain in Erenuman group differs from that in Placebo group; p = 0.96, ANOVA

2. Secondary Outcome: Change in SNOT-22 (Sino-nasal Outcome Test)
Description: The SNOT-22 consists of 22 items, each rated from 0 (no problem at all) to 5 (worst possible symptom). SNOT-22 total scores range from 0 to 110, with higher SNOT-22 total scores indicating worse symptoms. Reported as the change from baseline to six months.
Time Frame: Baseline, 1, 3 and 6 months
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 9 | 9
score on a scale | -10.1 (13.8) | -23.3 (25.2)
Statistical Analysis 1: Comparison: Erenumab vs Placebo; Test type: Equivalence — Test if the change in SNOT-22 score in Erenuman group differs from that in Placebo group; p = 0.19, ANOVA

3. Secondary Outcome: Change in Physical Function as Measured by Migraine Functional Impact Questionnaire (MFIQ)
Description: The MFIQ is a 26-item self-report questionnaire, developed to measure the subjective impact of migraine on physical functioning (everyday activities and physical impairment), as well as social and emotional functioning in the past seven days. The MFIQ Physical Function subscale is scored on a scale of 0-100, with higher scores indicating a greater impact. Reported as the change from baseline to six months.
Time Frame: Baseline, 1, 3 and 6 months
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 9 | 9
score on a scale | -3.3 (4.5) | -5.6 (6.5)
Statistical Analysis 1: Comparison: Erenumab vs Placebo; Test type: Equivalence — Test if the change in Physical Function as Measured by Migraine Function Impact in Erenuman group differs from that in Placebo group; p = 0.06, ANOVA

4. Secondary Outcome: Change in Usual Activities as Measured by Migraine Functional Impact Questionnaire (MFIQ)
Description: The MFIQ is a 26-item self-report questionnaire, developed to measure the subjective impact of migraine on physical functioning (everyday activities and physical impairment), as well as social and emotional functioning in the past seven days. The MFIQ usual activities subscale is scored on a scale of 0-100, with higher scores indicating a greater impact. Reported as the change from baseline to six months.
Time Frame: Baseline, 1, 3 and 6 months
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 9 | 9
score on a scale | -2.1 (4.4) | -10.9 (9.6)
Statistical Analysis 1: Comparison: Erenumab vs Placebo; Test type: Equivalence — Test if the change in Usual Activities as Measured by Migraine Function Impact in Erenuman group differs from that in Placebo group; p = 0.08, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Social Function as Measured by Migraine Function Impact Questionnaire (MFIQ)
Description: The MFIQ is a 26-item self-report questionnaire, developed to measure the subjective impact of migraine on physical functioning (everyday activities and physical impairment), as well as social and emotional functioning in the past seven days. The MFIQ Social Function subscale is scored on a scale of 0-100, with higher scores indicating a greater impact. Reported as the change from baseline to six months.
Time Frame: Baseline, 1, 3 and 6 months
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 9 | 9
score on a scale | -1.0 (3.6) | 5.7 (13.0)
Statistical Analysis 1: Comparison: Erenumab vs Placebo; Test type: Equivalence — Test if the change in Social Function as Measured by Migraine Function Impact in Erenuman group differs from that in Placebo group; p = 0.058, ANOVA

6. Secondary Outcome: Change in Emotional Function as Measured by Migraine Function Impact Questionnaire (MFIQ)
Description: The MFIQ is a 26-item self-report questionnaire, developed to measure the subjective impact of migraine on physical functioning (everyday activities and physical impairment), as well as social and emotional functioning in the past seven days. The MFIQ Emotional Function subscale is scored on a scale of 0-100, with higher scores indicating a greater impact. Reported as the change from baseline to six months.
Time Frame: Baseline, 1, 3 and 6 months
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 9 | 9
score on a scale | 0.4 (5.9) | -6.6 (5.7)
Statistical Analysis 1: Comparison: Erenumab vs Placebo; Test type: Equivalence — Test if the change in Emotional Function as Measured by Migraine Function Impact in Erenuman group differs from that in Placebo group; p = 0.02, ANOVA

7. Secondary Outcome: Change in Overall Impact (Global) as Measured by Migraine Function Impact Questionnaire (MFIQ)
Description: The MFIQ is a 26-item self-report questionnaire, developed to measure the subjective impact of migraine on physical functioning (everyday activities and physical impairment), as well as social and emotional functioning in the past seven days. The MFIQ Overall Impact is scored on a scale of 0-100, with higher scores indicating a greater impact. Reported as the change from baseline to six months.
Time Frame: Baseline, 1, 3 and 6 months
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 9 | 9
score on a scale | 0.11 (0.78) | -1.33 (1.00)
Statistical Analysis 1: Comparison: Erenumab vs Placebo; Test type: Equivalence — Test if the change in Overall Impact (global) as Measured by Migraine Function Impact in Erenuman group differs from that in Placebo group; p = 0.0036, ANOVA

8. Secondary Outcome: Change in Mean Number of Days Per Month With Significant Nasal Congestion
Description: Measured by daily diary completion via mobile app. Reported as the change from baseline to six months.
Time Frame: Baseline, 1, 3 and 6 months
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 13 | 12
days per month | -3.2 (6.0) | -2.8 (4.7)
Statistical Analysis 1: Comparison: Erenumab vs Placebo; Test type: Equivalence — Test if the change of average number of days per month with significant nasal congestion in Erenuman group differs from that in Placebo group; p = 0.83, ANOVA

9. Secondary Outcome: Change in Mean Number of Days Per Month With Significant Rhinorrhea
Description: Measured by daily diary completion via mobile app. Reported as the change from baseline to six months.
Time Frame: Baseline, 1, 3 and 6 months
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 13 | 12
days per month | -1.4 (5.7) | -1.8 (4.8)
Statistical Analysis 1: Comparison: Erenumab vs Placebo; Test type: Equivalence — Test if the change of average number of days per month with significant significant rhinorrhea in Erenuman group differs from that in Placebo group; p = 0.83, ANOVA

10. Secondary Outcome: Change in Mean Number of Days of Rescue Medication Used Per Month
Description: Measured by daily diary completion via mobile app. Reported as the change from baseline to six months.
Time Frame: Baseline, 1, 3 and 6 months
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 13 | 12
days per month | -5.2 (8.4) | -2.1 (3.8)
Statistical Analysis 1: Comparison: Erenumab vs Placebo; Test type: Equivalence — Test if the change in doses of rescue pain medications in Erenuman group differs from that in Placebo group; p = 0.35, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change From Baseline in Mean Daily Pain Score
Description: Measured by daily diary completion via mobile app on a scale of 1-10, where 1=no pain and 10=intense pain. Reported as the change from baseline to six months.
Time Frame: Baseline, 1, 3 and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erenumab | Placebo
Number analyzed (Participants) | 13 | 12
score on a scale | -0.9 (1.1) | -1.2 (1.6)
Statistical Analysis 1: Comparison: Erenumab vs Placebo; Test type: Equivalence — Test if the change from baseline in mean daily pain score in Erenuman group differs from that in Placebo group; p = 0.85, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Description: AEs and SAEs were systematically investigated at each study visit and self-reported and recorded using REDCap. Study team was notified via REDCap if subjects self-reported hypertension.
Arm/Group | Erenumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/13 | 0/12
Other Adverse Events (participants affected / at risk) | 7/13 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab (N=13) | Placebo (N=12)
Hypertension (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab (N=13) | Placebo (N=12)
Hypertension (Vascular disorders) | 6 | 4
Urinary tract infection (Renal and urinary disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Septoplasty (General disorders) | 0 | 1
Arm soreness/pain (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT04249427/Prot_SAP_000.pdf